CLINICAL TRIAL: NCT00559871
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Dose Response Study of the Efficacy, Safety and Tolerability of Fipamezole as an Oromucosal Fast Dissolving Tablet in the Treatment of Parkinson's Disease Patients.
Brief Title: Safety and Efficacy Study of Fipamezole in Treatment of Motor Dysfunctions in Parkinson's Disease
Acronym: Fjord
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juvantia Pharma Ltd (Industry)
Collaborators: Santhera Pharmaceuticals (Industry)
Responsible Party: Juha M. Savola, Director Clinical Development, Santhera Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-II-004
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Parkinson's Disease
Keywords: dyskinesia; movement disorders; basal ganglia diseases; JP-1730; Parkinson; end-of-dose wearing off; fluctuations
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Movement Disorders; Basal Ganglia Diseases | interventions — fipamezole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): One placebo tablet administered tid from Day 1 to 28
  Interventions: Drug: fipamezole
- 2 (Active Comparator): One 30-mg tablet of Fipamezole tid from Day 1 to 28
  Interventions: Drug: fipamezole
- 3 (Active Comparator): One 30-mg tablet of Fipamezole tid from Day 1 to 7; and one 60-mg tablet of Fipamezole tid from Day 8 to 28
  Interventions: Drug: fipamezole
- 4 (Active Comparator): One 30-mg tablet of Fipamezole tid from Day 1 to 7; one 60-mg tablet of Fipamezole tid from Day 8 to 14; and one 90-mg tablet of Fipamezole tid from Day 15 to 28
  Interventions: Drug: fipamezole

INTERVENTIONS:
Drug: fipamezole — Fipamezole in Zydis formulation three times per day for up to 28 days
  Other Names: JP-1730

SUMMARY:
The purpose of this study is to determine whether Fipamezole is effective in the treatment of levodopa-induced dyskinesia in advanced Parkinson's disease.

DETAILED DESCRIPTION:
This study is a multi-center, double-blind, placebo-controlled, multiple dose escalating, safety, tolerance, pharmacokinetics, and efficacy study of fipamezole administered in Parkinson's disease patients who are concomitantly being treated with a combination product of levodopa with a dopamine decarboxylase inhibitor (DDI) and possible other antiparkinson medication. Approximately 30 sites in the US and India will participate in this study. The patients will be randomized into one of four treatment arms to receive either fixed or ascending doses of Fipamezole (from 30 to 90 mg tid) or placebo. For efficacy assessments, levodopa-induced dyskinesia is assessed using a standardised rating scale. Time spent in 'Off' state or in 'On' state without dyskinesia, 'On' with non-troublesome dyskinesia or 'On' with troublesome dyskinesia, is assessed using patient diaries. Impact of dyskinesia on daily activities is quantified using a PDYS-26 questionnaire. To explore potential positive or negative impact of Fipamezole on cognitive functions, the study includes two cognitive tests. Finally, the study includes investigator assessments of CGI-I scales for dyskinesia, Parkinson's disease, and clinical condition in general.

ELIGIBILITY:
Main Inclusion Criteria:

* Idiopathic Parkinson's disease.
* Levodopa/DDI associated peak-dose dyskinesia which is at least moderately disabling and present for ≥25% of the waking day (UPDRS part IV, items 32 and 33, each ≥ 2).
* Stable Parkinson's medication for at least 1 month prior to randomization.
* Hoehn and Yahr Stages 1 to 4 during 'Off' period.
* Demonstrated ability to comprehend and give informed consent.
* Ability to complete patient diary.

Main Exclusion Criteria:

* Other clinically significant conditions apart from those typically associated with Parkinson's disease.
* Intake of medication associated with exacerbation of dyskinesia or with extrapyramidal side effects and tardive dyskinesia or induction of liver enzymes; neuroleptics; or specified drugs known to be substantially metabolized through the following cytochrome P450 isoenzymes: 1A2, 2B6, 2C19, 2C9, 2D6, and 2E1.
* Use of St. John's Wort or Ginkgo Biloba within 48 hrs prior to randomization and until the last treatment day with the study medication.
* Intake of an investigational drug within 30 days prior to initial screening.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of 3 different doses of fipamezole with that of placebo on dyskinesia as assessed by a dyskinesia assessment scale. | 28-days treatment

SECONDARY OUTCOMES:
To compare efficacy of 3 different doses of fipamezole with that of placebo on the mean daily 'Off' time, as recorded in the patient diary. | 28-days treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. LeWitt, M.D., Principal Investigator — Henry Ford Health Systems, Franklin Pointe Medical Center
Locations (36):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Neurology Clinic PC, Northport, Alabama
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Parkinson and Movement Disorder Institute, Fountain Valley, California
  - University of California Irvine, Irvine, California
  - Coastal Neurological Medicine Group, La Jolla, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Parkinson's Disease and Movement Disorder Center, Boca Raton, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Pharmax Research Clinic, Miami, Florida
  - University of Miami, Miami, Florida
  - Collier Neurological Clinic, Naples, Florida
  - University of South Florida, Parkinson's Disease and Movement Center, Tampa, Florida
  - Emory Healthcare, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Parkinson Disease Center - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maryland Parkinson's Disease and Movement Disorder Center, Baltimore, Maryland
  - U Mass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Health Systems, Franklin Pointe Medical Center, Southfield, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - Neurology Group of Bergen County, Ridgewood, New Jersey
  - Biomedical Research Alliance of New York, Forest Hills, New York
  - Duke Health Center at Morreene Road, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Semmes Murphey Neurologic and Spine Institute, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Neurology Associates, San Antonio, Texas
- India (7):
  - Max Superspecialty Hospital, Saket, New Delhi
  - Neurology centre, Ahmedabad
  - St John's Medical College & Hospital, Bangalore
  - M S Ramaiah Medical College Hospital, Bangalore
  - Nizam's Institute of Medical Sciences, Hyderabaad
  - Chatrapati Sahuji Maharaj Medical University, Lucknow
  - J.S.S. Medical College and Hospital, Mysore